CLINICAL TRIAL: NCT04732520
Title: The Galvanize Therapeutics Early Stage, Non-Small Cell Lung Cancer, Treat and Resect Study
Brief Title: Feasibility Study of the Aliya System in the Treatment of Early Stage Non-small Cell Lung Cancer
Acronym: INCITE ES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galvanize Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-00009
Record Dates: First submitted 2021-01-28; First posted 2021-02-01 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental): Patients participating in the treatment group will undergo pulsed electric field (PEF) treatment of a single NSCLC nodule measuring 1 to 4 cm by CT, using the Aliya System. The treatment may be performed endoluminally in conjunction with a diagnostic bronchoscopy, or percutaneously.
  Interventions: Device: Pulsed electric field treatment using the Aliya System
- Control (No Intervention): Patients declining to participate in the treatment arm may self-select to participate in an observational control arm.

INTERVENTIONS:
Device: Pulsed electric field treatment using the Aliya System — pulsed electric field treatment of a single NSCLC tumor
  Arms: Treatment

SUMMARY:
A prospective, two-arm, non-randomized, concurrently controlled, multi-center, open-label, treat and resect study following patients to 1 year. The study is designed to evaluate the safety and feasibility of the Aliya System for the ablation of solid tumors using pulsed electric field (PEF) energy delivery. The study is intended for adult patients with suspected or confirmed NSCLC 8th ed. Stage IA2, IA3 or IB (>1 to ≤4 cm solitary lesion) who are surgical candidates and have not received treatment for the index tumor in the last two years.

DETAILED DESCRIPTION:
This study is to evaluate the safety and initial feasibility of Pulsed Electric Field (PEF) treatment of NSCLC tumors prior to surgical resection.

Treatment may be delivered via either an endoluminal (bronchoscopic) or percutaneous approach at the discretion of the clinical investigator utilizing two available device configurations:

* Endoluminal: Galvanize Aliya System with commercially available TBNA Needle (e.g., PeriView FLEX) and RF probe electrode
* Percutaneous: Galvanize Aliya System with compatible commercially available RF needle and RF probe electrode

The study will enroll and treat up to 30 adult patients with early stage NSCLC at up to 5 clinical sites. Patients meeting all eligibility criteria who elect not to undergo the PEF treatment will be offered the opportunity to participate in a concurrent control arm. Up to 10 patients will be included in the control group. A total of up to 40 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of solitary NSCLC nodule 8th ed. stage IA2, IA3 or IB
* Nodule measuring > 1 cm and ≤4 cm diameter by CT size estimate (e.g. T1b, T1c, T2a), with a minimum 1 cm solid component
* High pre-procedure probability of malignancy as determined by the investigator
* Patient has been evaluated by a thoracic surgeon and deemed a candidate for definitive lung tissue resection
* Patient is, in the opinion of the principal investigator, able to adhere to and undergo bronchoscopy, surgical procedure and post-treatment care

Exclusion Criteria:

* Additional pulmonary nodules requiring intervention
* Patient is receiving concurrent cancer treatment (e.g. external beam radiation therapy, brachytherapy, chemotherapy, targeted therapy, immunotherapy, other focal therapy) or has received treatment for the index tumor in the last two years
* Patient has implanted lung devices or electronic devices
* Patient has N1 disease
* Patient is immune compromised or receiving immune modulating medication
* Recurrent NSCLC within 2 years of initial definitive treatment
* Previous checkpoint inhibitor treatment for another cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Device and Procedure related serious adverse event rate | 30 days
  The rate of system-related and procedure-related serous adverse events (SAEs)

SECONDARY OUTCOMES:
Technical Success rate | Acute procedure
  The frequency with which the clinician can access the index tumor and delivery energy

CONTACTS AND LOCATIONS:
Locations (4):
- Prince of Wales Hospital, Shatin, Hong Kong
- Radboud University Medical Center, Nijmegen, Netherlands
- Spain (2):
  - Fundacion Instituto de Investigation Sanitaria de la Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario de Salamanca, Salamanca